CLINICAL TRIAL: NCT03385213
Title: Structural of the Gut Mucosal Microbiota is Associated With Colorectal Cancer Relapses After Curative Surgery
Brief Title: Gut Mucosal Microbiota is Associated With Colorectal Cancer Relapse
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Yunwei Wei 2017 -2
Record Dates: First submitted 2017-12-17; First posted 2017-12-28 (Actual); Last update posted 2018-05-09 (Actual); Status verified 2017-12

CONDITIONS: Gut Microbiota; Colorectal Cancer
Keywords: Microbiota; colorectal cancer; relapse; surveillance
MeSH Terms: conditions — Colorectal Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Human fecal and gut mucosal samples for DNA extraction
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Relapse: Patients who suffered colorectal cancer relapse after curative surgery
- Remission: Patients who get remission after curative surgery

SUMMARY:
Colonic microbiome has been found to contribute to the development of colorectal cancer. We speculate that gut microbiota related to colorectal cancer relapse after curative treatment. This study aim to discover if any difference of gut microbiota exist in patients who suffer from cancer relapse compared with patients who do not. Finally develop patient-centred programmes of surveillance protocols base on microbiota analysis.

DETAILED DESCRIPTION:
Treatments for colorectal cancer of all stages have evolved considerably over the past two decades, resulting in improved long-term outcomes. After curative treatment, however, 30% of patients with stage I-III and up to 65% of patients with stage IV colorectal cancer develop recurrent disease.

The human colon plays host to a diverse and metabolically complex community of microorganisms. While the colonic microbiome has been found to contribute to the development of colorectal cancer. Investigators speculate that gut microbiota related to colorectal cancer relapse after curative treatment.

Patients are routinely offered surveillance in order to detect disease recurrence at an early, asymptomatic stage, with the intention of improving survival. Nevertheless, controversy continues to surround the optimal surveillance protocols. Investigators aim to discover if any difference of gut microbiota is exist in patients who suffer from relapse compared with patients who do not.

Future surveillance after colorectal cancer treatment should focus on risk-stratification and should incorporate current knowledge on risk of recurrence in relation to the biology of the tumour as well as gut microbiota feature. Finally investigators will develop patient-centred programmes of surveillance protocols base on microbiota analysis.

ELIGIBILITY:
Inclusion Criteria:

* Requirements of informed consent and assent of participant, parent or legal guardian as applicable
* Patients with colorectal cancer scheduled for radical coloproctectomy and between the age of 18 and 75 years old without considering sex.
* Patients with BMI= 18.5-23.9
* Participants can follow the visit plan

Exclusion Criteria:

* Patients with colorectal cancer with distant metastasis
* Chronic renal diseases and hepatic cirrhosis
* Chronic ischemic heart disease with unstable angina, chronic heart failure at class III or IV and acute myocardial infarction in the last 6 months
* Individuals with a history of Chronic diarrhea
* Individuals with a history of Diabetes mellitus
* Individuals with a history of Hypertension
* Individuals with a history of autoimmune diseases
* Use of antibiotics and probiotics 3 mouth before samples collection
* Individuals with a history of abdominal operation due to any reason
* Individuals with any history of cancer other than colorectal cancer
* Individuals with Inflammatory bowel disease

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colorectal cancer is a major cause of cancerrelated deaths and the third most commonly diagnosed cancer worldwide. After curative treatment, however, 30% of patients with stage I-III and up to 65% of patients with stage IV CRC develop recurrent disease.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-05-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Transcriptional changes in gut microbiota | Baseline, 6 months after surgery, 12 months after surgery, 24 months after surgery
  16S rRNA gene sequencing will be performed with stander procedure

SECONDARY OUTCOMES:
Epigenetic changes | Baseline, 6 months after surgery, 12 months after surgery, 24 months after surgery
  DNA methylation levels are analysed at baseline and after probiotics use in tissue samples

CONTACTS AND LOCATIONS:
Overall Officials: Yunwei Wei, Study Director — First Affiliated Hospital of Harbin Medical University
Locations (1):
- Yunwei Wei, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No